CLINICAL TRIAL: NCT03457389
Title: Comparison of Treatment Outcome of Cabergoline According to Target Prolactin Levels in Patients With Prolactinoma: A Prospective, Randomized, Open Label, Active-controlled, Clinical Trial
Brief Title: Comparison of Treatment Outcome of Cabergoline According to Target Prolactin Levels in Patients With Prolactinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Hee Kim, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1711-119-901
Record Dates: First submitted 2018-01-23; First posted 2018-03-07 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-09

CONDITIONS: Pituitary Adenoma; Prolactinoma; Pituitary Tumor; Recurrence Tumor
Keywords: Prolactinoma; Cabergoline; Recurrence
MeSH Terms: conditions — Pituitary Neoplasms; Prolactinoma; Recurrence | interventions — Cabergoline

STUDY DESIGN:
Intervention Model Description: One experimental group and one control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Serum prolactin level is adjusted to less than 5 ng/mL during cabergoline administration.
  Interventions: Drug: Cabergoline
- Control group (Active Comparator): Serum prolactin level is adjusted to normal range during cabergoline administration.
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline — Cabergoline tablet
  Other Names: Caverlactin

SUMMARY:
The aim of this study is to investigate whether inhibition of serum prolactin levels below normal range during cabergoline administration may reduce the recurrence rate after drug withdrawal in patients with prolactinomas.

DETAILED DESCRIPTION:
Prolactinoma patients will be assigned to a experimental group that maintains serum prolactin levels below 5 ng/mL and a control group that maintains normal serum prolactin levels. After that, cabergoline will be maintained at a therapeutic dose for 130 weeks. After cabergoline is discontinued, patients will be followed up with serum prolactin measurement for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults, male or female aged 19 years or older
* diagnosed with prolactinoma
* No previous history of surgery, medication, or radiation therapy

Exclusion Criteria:

* Invasive prolactinomas except invading cavernous sinus
* Taking dopaminergic medications
* Taking medications that can affect serum prolactin level (including estrogenic hormone, oral contraceptive drugs, intrauterine devices)
* Hyperprolactinemia due to secondary causes
* History of pituitary apoplexy within the last 3 months
* Patients with mental illness that should avoid dopamine agonists
* Patients with history of cardiac valve diseases
* Patients with history of pulmonary fibrosis, retroperitoneal fibrosis, and cystic fibrosis
* Moderate degree of hepatic or renal insufficiency (IDMS Modification of Diet in Renal Disease glomerular filtration rate (MDRD GFR) <45 ml/min/1.73m2)
* Patients with cabergoline hypersensitivity reaction
* Pregnant or breast feeding patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate within 1 year after cabergoline withdrawal | From 4 year to 5 years after cabergoline administration
  Record of PRL levels on every 3 month follow-up visit

SECONDARY OUTCOMES:
Time to normalization of serum prolactin level | Up to 1 year
  Record of PRL levels on follow-up visit
Change from baseline on tumor volume measured by pituitary MRI | Up to 3 years
  Record of he tumor volume from pituitary MRI on every 12-month follow-up visit
Change from baseline of visual field defect | Up to 3 years
  Record the Visual field scale on every 6 month follow-up visit,

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Kim, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No